CLINICAL TRIAL: NCT02419456
Title: Phase 1 Pharmacokinetic Trial of Two Intravaginal Rings (IVRs) Containing Different Dose Strengths of Vicriviroc (MK-4176) and MK-2048
Brief Title: Pharmacokinetics of Two Intravaginal Rings (IVRs) Containing Different Dose Strengths of Vicriviroc (MK-4176) and MK-2048
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTN-028; 12022 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2016-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MK-2048A Intravaginal Ring (IVR) (Low Dose) (Experimental): The MK-2048A IVR (Low Dose) will be inserted during the enrollment visit (Day 0), and it will be removed on Day 28.
  Interventions: Drug: MK-2048A IVR (Low Dose)
- MK-2048A IVR (Original Dose) (Experimental): The MK-2048A IVR (Original Dose) will be inserted during the enrollment visit (Day 0), and it will be removed on Day 28.
  Interventions: Drug: MK-2048A IVR (Original Dose)

INTERVENTIONS:
Drug: MK-2048A IVR (Low Dose) — Contains 91 mg of vicriviroc (MK-4176) and 10 mg of MK-2048.
  Arms: MK-2048A Intravaginal Ring (IVR) (Low Dose)
Drug: MK-2048A IVR (Original Dose) — Contains 182 mg of vicriviroc (MK-4176) and 30 mg of MK-2048.
  Arms: MK-2048A IVR (Original Dose)

SUMMARY:
Intravaginal rings (IVRs) may offer an ideal way to deliver antiretroviral (ARV) drugs to prevent HIV infection. This study will evaluate the pharmacokinetics and safety of two IVRs containing different doses of a combination of two HIV ARV drugs, vicriviroc (VCV) (MK-4176) and MK-2048, in healthy, HIV-uninfected women.

DETAILED DESCRIPTION:
The development of safe and effective HIV prevention strategies remains a global health priority. IVRs are currently being studied as a method to deliver HIV ARV drugs in women. This study will evaluate the pharmacokinetics and safety of two IVRs containing different doses of a combination of two HIV ARV drugs, vicriviroc (VCV) (MK-4176) and MK-2048, in healthy, HIV-uninfected women.

This study will enroll healthy, HIV-uninfected women, 18 to 45 years old. Participants will be randomly assigned to receive either the low dose MK-2048A IVR or the original dose MK-2048A IVR. Participants will receive their assigned IVR at the enrollment visit, and the IVR will be removed on Day 28. Participants will attend study visits at screening, enrollment (Day 0), and Days 1, 2, 3, 7, 14, 21, 28, 29, 30, 31, and 35. Study visits may include medical history reviews, physical examinations, blood collection, pelvic specimen collection, urine collection, and counseling and adherence assessments.

ELIGIBILITY:
Inclusion Criteria:

* Born female. Note: Participants who were female at birth, who now identify as male, will not be excluded so long as they are not on female-to-male transition therapy.
* Age 18 through 45 years (inclusive) at screening, verified per site SOPs (standard operating procedures)
* Able and willing to provide written informed consent to be screened for and take part in this study (MTN-028)
* Able and willing to provide adequate locator information, as defined by the site SOPs
* HIV-uninfected, based on testing performed by study staff at screening and enrollment (per applicable algorithm in Appendix II of the protocol) and willing to receive results
* In general good health at screening and enrollment, as determined by the site Investigator of Record (IoR) or designee
* At screening, participant states willingness to abstain from receptive sexual activity (including penile-vaginal intercourse, anal intercourse, receptive oral intercourse, finger stimulation, and the use of sex toys) for the 5 days prior to the enrollment visit and for the duration of study participation
* Per participant report, using an effective method of contraception at enrollment, and intending to continue the use of an effective method for the duration of study participation. Effective methods for MTN-028 include: hormonal methods (except contraceptive IVRs), intrauterine device (IUD) inserted at least 28 days prior to enrollment, engages in sex exclusively with women, sterilized (self or partner), and/or sexually abstinent for the past 90 days
* Women over the age of 21 (inclusive) must have documentation of a satisfactory Pap within the past 3 years prior to enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result. If otherwise eligible women do not have documentation of a recent Pap test, one may be performed at the screening visit.
* Per participant report at screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products for the duration of study participation
* Per participant report at screening, regular menstrual cycles with at least 21 days between menses. Note: This criterion is not applicable to participants who report using a progestin-only method of contraception at screening (e.g., Depo-Provera or levonorgestrel-releasing IUD) nor to participants using continuous combination oral contraceptive pills, as the absence of regular menstrual cycles is an expected, normal consequence in this context.
* At screening, participant states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina, including but not limited to, spermicides, female condoms, diaphragms, contraceptive IVRs, vaginal medications, menstrual cups, cervical caps (or any other vaginal barrier method), douches, lubricants, sex toys (vibrators, dildos, etc.) for the 5 days prior to enrollment and for the duration of their study participation

Exclusion Criteria:

* Participant report of any of the following at screening or enrollment:

  * History of adverse reactions to any of the components of the study products
  * Non-therapeutic injection drug use in the 12 months prior to screening and enrollment
  * Post-exposure prophylaxis (PEP) for HIV exposure within 6 months prior to enrollment
  * Pre-exposure prophylaxis (PrEP) for HIV prevention within the 6 months prior to enrollment
  * Regular use and/or anticipated regular use during the period of study participation of CYP3A inducer(s) and/or inhibitor(s)
  * Use and/or anticipated use during the period of study participation of female-to-male transition therapy
  * Chronic and/or recurrent candidiasis
  * Gonorrhea, chlamydia and/or syphilis diagnosis in the 6 months prior to enrollment
  * Last pregnancy outcome 90 days or less prior to screening
  * Currently breastfeeding
  * Has had a hysterectomy
  * Intends to become pregnant within the next 3 months
  * Has plans to relocate away from the study site area in the next 3 months
  * Current sexual partner is known to be HIV-positive at screening or enrollment
* Reports participating in any other research study involving drugs, medical devices, or vaginal products within 60 days or less prior to enrollment
* At screening or enrollment, as determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease
* Has any of the following laboratory abnormalities at screening:

  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher
  * Calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula, where creatinine clearance (female) in mL/min = (140 - age in years) x (weight in kg) x (0.85)/72 x (creatinine in mg/dL)
  * Hemoglobin Grade 1 or higher
  * Platelet count Grade 1 or higher
  * White blood count Grade 2 or higher
  * Positive hepatitis B surface antigen (HBsAg) test result
  * Positive anti-hepatitis C virus (HCV) test result
  * International normalized ratio (INR) greater than 1.5 × the site laboratory upper limit of normal (ULN)
  * Note: Otherwise eligible participants with an exclusionary test result (other than HIV, hepatitis B virus [HBV], or HCV) can be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
* Pregnant at either screening or enrollment. Note: A documented negative pregnancy test performed by study staff is required for inclusion; however a self-reported pregnancy is adequate for exclusion from screening/enrollment into the study.
* Diagnosed with urinary tract infection (UTI) at screening or enrollment. Note: Otherwise eligible participants diagnosed with UTI during screening will be offered treatment. If within the 45 day screening window treatment is complete and symptoms have resolved the participant may be enrolled.
* Diagnosed with pelvic inflammatory disease, reproductive tract infection (RTI) or a sexually transmitted infection (STI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment/) at screening or enrollment. Note: With the exception of gonorrhea, chlamydia and/or syphilis, otherwise eligible participants diagnosed with a RTI during screening will be offered treatment. If within the 45 day screening window treatment is complete and symptoms have resolved, the participant may be enrolled.
* At enrollment, has a clinically apparent Grade 1 or higher pelvic exam finding (observed by study clinician or designee) per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), Addendum 1, Female Genital Grading Table for Use in Microbicide Studies. Note: Cervical friability bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.
* At screening, severe pelvic relaxation such that either the vaginal walls or the uterine cervix descend beyond the vaginal introitus with valsalva maneuver or has pelvic anatomy that compromises the ability to adequately assess vaginal safety
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessment of vaginal fluid concentrations of MK-4176 and MK-2048 during and after IVR use | Measured through Day 35
Assessment of blood plasma concentrations of MK-4176 and MK-2048 during and after IVR use | Measured through Day 35
Assessment of cervical tissue concentrations of MK-4176 and MK-2048 during and after IVR use | Measured through Day 35
Number of genitourinary events Grade 1 or higher judged to be related to study product | Measured through Day 35
  As defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009), Addendum 1, (Female Genital Grading Table for Use in Microbicide Studies)
Number of adverse events Grade 2 or higher | Measured through Day 35
  As defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009)

SECONDARY OUTCOMES:
Measurement of residual drug levels in IVRs | Measured through Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, MD, MPH, Study Chair — San Francisco Department of Public Health
Locations (1):
- Bridge HIV CRS, San Francisco, California, United States

REFERENCES:
- [Derived] Liu AY, Zhang J, Anderson PL, Wagner T, Pan Z, Peda M, Gomez K, Beamer M, Jacobson C, Strizki J, Dezzutti CS, Piper JM; MTN-028 Protocol Team for the Microbicide Trials Network. Phase 1 Pharmacokinetic Trial of 2 Intravaginal Rings Containing Different Dose Strengths of Vicriviroc (MK-4176) and MK-2048. Clin Infect Dis. 2019 Mar 19;68(7):1129-1135. doi: 10.1093/cid/ciy652. PMID 30289444